CLINICAL TRIAL: NCT02237378
Title: Evaluation of Cardiopulmonary Metabolism and Pulmonary Vascular Remodeling in Pulmonary Hypertension Associated With Left Heart Disease
Brief Title: A Pilot Study Evaluating Heart and Lung Metabolism in Pulmonary Hypertension Associated With Left Heart Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrolment
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20140602
Record Dates: First submitted 2014-08-29; First posted 2014-09-11 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Hypertension
Keywords: FDG lung and RV uptake
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG PET scan (Experimental): A PET scan using F-18 FDG, N-13 Ammonia will be performed
  Interventions: Radiation: FDG PET scan

INTERVENTIONS:
Radiation: FDG PET scan — Following an overnight fast, subjects will be positioned in the Discovery 660 PET/VCT scanner. Following a scout scan to confirm patient positioning, low dose xray CT scan is performed for photon attenuation. A 20 minute dynamic PET scan is started simultaneously with 3 MBq/kg of N-13 ammonia to measure myocardial perfusion. Following N-13 decay,a 60 minute dynamic PET scan with 3 MBq/kg F-18- FDG to measure myocardial glucose uptake. Blood sampling for glucose and insulin will occur at pre specified time points throughout the scan.
  Other Names: F-18-FDG; N-13 ammonia

SUMMARY:
Right ventricular (RV) failure is the leading cause of death in pulmonary arterial hypertension. (PAH) Right ventricular ejection fraction is one of the most important predictors of prognosis in heart failure patients regardless of cause. It is estimated that 30-50% of patients with heart failure and preserved ejection fraction (HFpEF) have right ventricular dysfunction and up to 70% of these patients will have significant pulmonary hypertension (PH), both of which are related to much worse prognosis. Right ventricular failure is becoming an increasingly prevalent and significant cause of morbidity in patients with left heart disease. Despite the significance of RV function to survival, there are no therapies available that directly or selectively improve RV function.

The overall theme of this research project is to evaluate the mechanisms that contribute to the cause of right heart failure. This small study is designed to look at the role of heart and lung metabolism and pulmonary hypertension as they relate to the development of right heart failure in cardiovascular disease.(PH-LHD)

DETAILED DESCRIPTION:
The hemodynamic definition of PH-LHD involves a mean pulmonary artery pressure (mPAP) >25mm Hg at rest and pulmonary capillary wedge pressure (PCWP) of ≥15.The coexistence of mitral insufficiency is also a characteristic of PH-LHD. HFpEF is a condition caused by impaired relaxation of a stiffened myocardium as a consequence of an increased load to the left ventricle due to elevated systemic pressures.

Pulmonary hemodynamics can be used to classify PH LHD as either passive or reactive, irrespective of LV function. It has been suggested that diastolic pressure gradient (DPG) may offer added prognostic value as a more accurate indicator of pulmonary vascular remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide their written informed consent to participate in the study after having received adequate previous information and prior to any study specific procedures.
* At least 18 years of age at the time of screening.
* Patients with PH secondary to left heart disease (known as group II PH) defined as a mean PAP>25 mmHg and a PCWP of ≥15 mmHg.

Exclusion Criteria:

* All other types of pulmonary hypertension including Dana Point Classification Group 1, 3, 5.
* Type II Diabetes mellitus requiring medical therapy
* Previous myocardial infarction within the 3 months prior to screening.
* Renal insufficiency (glomerular filtration rate < 30 ml/min.
* ALT or AST > 3times ULN and/or severe hepatic insufficiency.
* Contraindication to MRI imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cardiac and pulmonary metabolism role in development of right heart failure in pulmonary hypertension in left heart disease. | Baseline
  Relationship between lung fludeoxyglucose (FDG)uptake and hemodynamic type pulmonary hypertension using PET scanning

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Mielniczuk, MD, Principal Investigator — University of Ottawa Heart Institiute
Locations (1):
- University of OttawaHeart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only 2 participants were enrolled in this study. One of the main reasons was no clinical indication to repeat a right heart catherization in this population.